CLINICAL TRIAL: NCT04423419
Title: the Efficacy of Peri-articular Nerve Group Block(PENG Block)Versus Fascia Iliaca Block on Immediate Post Operative Pain and Opioid Consumption After Hip Arthroscopy
Brief Title: Peri-articular Nerve Group Block Versus Fascia Iliaca Block on Postoperative Pain After Hip Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safa Sayed Noaman, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: postoperative pain
Record Dates: First submitted 2020-05-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Analgesia
Keywords: post operative pain; hip arthroscopy
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: group A will undergo PENG block group B will undergo fascia iliaca block groupC will receive iv analgesia
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient and the assessor will mask about type of block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Other): will undergo Peri -articular nerve group block for hip joint under ultrasound guide as analgesia post operative after hip arthroscopy
  Interventions: Procedure: PENG block
- B (Other): will undergo ultrasound guided fascia iliaca block as postoperative analgesia after hip arthroscopy
  Interventions: Procedure: fascia iliaca block
- C (Other): will receive ordinary IV analgesia during operation hip arthroscopy
  Interventions: Other: IV analgesia

INTERVENTIONS:
Procedure: PENG block — The US probe placed in a transverse plane over the AIIS . the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 80-mm needle was inserted from lateral to medial to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic drug was injected while observing for adequate fluid spread for a total volume of 20 mL of Bupivacain 0.25%
  Other Names: injection of local anasthetics drug in peri-articular nerves of hip joint
  Arms: A
Procedure: fascia iliaca block — ultrasound guidance landmarks are the anterior superior iliac spine and the pubic tubercle (inguinal ligament). The injection site along the lateral one-third of aline joining the anterior superior iliac spine (ASIS) and pubic tubercle (PT) targeting the compartment between fascia iliaca and fascia lata ,the total volume of injection is 20ml of Bupivacain 0.25%
  Other Names: injection of local anathetics drug in fascia ilica space
  Arms: B
Other: IV analgesia — IV analgesia
  Other Names: no block
  Arms: C

SUMMARY:
The study aims to evaluate the efficacy of pericapsular nerve group block versus fascia iliaca block in reducing post operative pain within the first 24 hours following hip arthroscopy

DETAILED DESCRIPTION:
In recent decades hip arthroscopy gained popularity and the number of procedures increase every year , due to the widening range of indications, as femoroacetabular impingement, labral tears, chondral injuries, loose bodies, osteonecrosis and septic arthritis Pain after hip arthroscopy due to several factors. divided in two regions. First the intra-articular where pain originates from the joint capsule (capsulotomy), a repaired labrum or bony resection. Outside the joint caused by traction, the portal tracts and extravasation of irrigation , soft tissue swelling.

the hip joint found to be innervated from the femoral nerve for its anterior part, the obturator nerve for its antero-medial part, the sciatic nerve for its posterior part, and the nerve to the quadratus femoris muscle for its postero-medial par

Pericapsular Nerve Group (PENG) Block aims to block the articular branches of the accessory obturator and femoral nerve Also, it could spread to block the obturator nerve and its articular branches the high articular branches from FN and AON are found between the anterior inferior iliac spine(AIIS) and the ilio pubic eminence (IPE), whereas the ON is located close to the inferomedial acetabulum.

The fascia iliaca compartment is a virtual space anteriorly limited by the posterior surface of the fascia iliaca, posteriorly by the iliacus muscle and is cranially in continuation with the space between quadratus lumborum muscle and its fascia . Three important nerves for hip innervation are located in this space, the femoral nerve, obturator nerve and lateral femoral cutaneous nerve

ELIGIBILITY:
Inclusion Criteria:

age 16-60 years old ASA physical status I or II scheduled for hip arthroscopy

Exclusion Criteria:

* pregnancy or breast feeding
* neurological deficits or neuropathy
* opioid addict
* local skin infections, bleeding diathesis, and coagulopathy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficacy of pericapsular nerve group block versus fascia iliaca block in reducing post operative pain within the first 24 hours following hip arthroscopy | 24 hours
  by question the patient about pain and its degree using visual analogue pain score( VAS score),it takes score from (0-10) according to severity of pain ,higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
duration of the analgesic effect of the block | 24 hours
  evaluate duration of the analgesic effect of the block by calculating The time passed from block to the patient first analgesia request and total cumulative doses of analgesia

CONTACTS AND LOCATIONS:
Overall Officials: essam sharkawy, lecturer, Study Director — Assiut University

REFERENCES:
- [Background] 1_ Colvin AC, Harrast J, Harner C. Trends in hip arthroscopy. J Bone Joint Surg Am 2012; 94: e23. 2_ Tan CO, Chong YM, Tran P et al. Surgical predictors of acute postoperative pain after hip arthroscopy. BMC Anesthesiol 2015; 15:96. 3- Jerry G. Xing,*yMD, MSc, FRCSC, Faraj W. Abdallah,zMD, Richard Brull,§MD, FRCPC,Stephanie Oldfield,§Andrew Dold,yMD, M. Lucas Murnaghan,||MD, MEd, FRCSC,and Daniel B. Whelan,{MD, FRCSC Preoperative Femoral Nerve Block for Hip Arthroscopy Randomized, Triple-Masked Controlled Trial The American Journal of Sports Medicine 2015 4_, Gardner E. The innervation of the hip joint. Anat Rec. 1948;101:353-371. 5_ Girón-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular nerve group (PENG) block for hip fracture. RegAnesth Pain Med. 2018; 43(8):859-63. 6_ Bhatia A, Hoydonckx Y, Peng P, Cohen SP. Radiofrequency procedures to relieve chronic hip pain. An evidence-based narrative review. Reg Anesth Pain Med. 2018;43:72-83. 7_S.M.White,R.Griffiths,J.Holloway,andA.Shannon,"AnaesthesiaforproximalfemoralfractureintheUK:firstreportfrom theNHShipfractureanaesthesianetwork,"Anaesthesia,vol.65, no.3,pp.243-248,2010.